CLINICAL TRIAL: NCT06109623
Title: Study on the Correlation Between Changes in Steroid Hormone Levels and Stress Urinary Incontinence in Women
Brief Title: Correlation Between Changes in Sex Hormone Levels and Stress Urinary Incontinence in Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Chun-Wu Pan, Professor, RenJi Hospital
Other Study IDs: IIT-2023-0135
Record Dates: First submitted 2023-10-10; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Urinary Incontinence,Stress
Keywords: Stress Urinary Incontinence; Steroid Hormone; Case-Control Study
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Observation; Gonadal Steroid Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SUI group: Female patients diagnosed with stress urinary incontinence in our hospital, who met the inclusion and exclusion criteria, and received six sex hormone tests.
  Interventions: Other: observation; Other: sex hormone
- control group: Patients with non-stress urinary incontinence
  Interventions: Other: observation; Other: sex hormone

INTERVENTIONS:
Other: observation — To observe the changes and differences of steroid hormones between stress urinary incontinence group and control group.
Other: sex hormone — Six indicators of steroid hormones (estrogen, testosterone, follicle stimulating hormone, luteinizing hormone, pituitary prolactin, progesterone)

SUMMARY:
The goal of this observational study is to learn about the relationship between stress urinary incontinence and endogenous steroids in women, especially its occurrence and severity with androgens and estrogens. The main questions it aims to answer are:

* Association between stress urinary incontinence and endogenous steroids in women
* Risk factors associated with stress urinary incontinence in women Participants will be asked to provide basic clinical information as well as results of measurements of serum steroid hormone levels.

Researchers will compare Stress urinary incontinence group and control group to see if the changes of sex hormone levels were statistically significant.

DETAILED DESCRIPTION:
By comparing the differences of six hormones between female patients with stress urinary incontinence (SUI) and non-SUI patients (patients without pelvic floor muscle dysfunction and lower urinary tract dysfunction) aged ≥20 years, especially the changes of androgen and estrogen levels, the correlation between the changes of hormone levels and stress urinary incontinence was obtained. Multivariate logistic regression analysis was used to analyze the relationship between hormones and urinary incontinence, and further correlation analysis was performed for statistically significant hormones. Estrogen and androgen were divided into four groups: normal estrogen/normal androgen group, decreased estrogen/normal androgen group, normal estrogen/decreased androgen group, decreased estrogen/decreased androgen group. Stratified analysis was performed to analyze whether there was an interaction between the two hormones and exclude confounding effects. Finally, the data were further analyzed by sensitivity analysis of baseline characteristics, and the known risk factors were verified in this trial, including age, parity, menopausal status, genetic factors, obesity, and on this basis, the correlation between pelvic surgery history, diabetes, hypertension, smoking and stress urinary incontinence was explored.

ELIGIBILITY:
Inclusion Criteria:

- Experimental Group

1. women aged ≥20 years
2. Stress urinary incontinence diagnosed in our hospital;
3. Six hormone tests were performed in our hospital; Control group

(1) women aged ≥20 years; (2) diseases other than stress urinary incontinence diagnosed by our hospital; (2) Six hormone tests were performed in our hospital;

Exclusion Criteria:

1. Pelvic organ prolapse, overactive bladder, urge urinary incontinence, overflow urinary incontinence, mixed urinary incontinence;
2. patients who received hormone replacement therapy within 6 months;
3. estrogen-dependent diseases, such as endometriosis, uterine leiomyoma, ovarian tumors;
4. the presence of gynecological malignant tumors or other diseases affecting hormone secretion;
5. the presence of nervous system diseases.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients aged ≥20 years with stress urinary incontinence and patients without stress urinary incontinence. Both inclusion and exclusion criteria were met.
Sampling Method: Non-Probability Sample
Enrollment: 1226 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Baseline characteristics | baseline, pre-procedure
  The results of this study were described by statistical methods. Descriptive statistical analysis was performed on the baseline characteristics of patients in the SUI group and the control group. Categorical variables were described by frequency (%), and Pearson chi-square test or Fisher Exact test was used. Continuous variables describe their mean (SD) or median data (interquartile range) according to their normality, and comparisons between groups were performed using the independent t-test (normal) or Mann Whitney test (non-normal).
Association analysis between stress urinary incontinence and androgen levels | immediately after the procedure
  The association between stress urinary incontinence and the lowest quartile of serum testosterone was examined by a weighted, multivariate logistic regression model. Odds ratios and 95% confidence intervals were calculated for each outcome of interest. All models were adjusted for age, BMI, parity, menopausal status, history of pelvic surgery, hypertension, and diabetes. Two-sided p values of 0.05 or less were considered to indicate statistical significance.

SECONDARY OUTCOMES:
Sensitivity analysis or stratified analysis | through study completion, an average of 6 month
  The association between hormone levels and stress urinary incontinence is affected by many uncertain factors, such as population characteristics and disease history. In order to avoid bias of results caused by uncertain factors, sensitivity analysis or stratified analysis of these factors is required. This project planned to perform sensitivity or stratified analyses by grouping the subjects into multiple subgroups (grouped by age, history of childbirth, history of hypertension, history of diabetes, history of pelvic surgery, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Wu Pan, professor, Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University,

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the primary results of the trial, including data on the primary and secondary end points, after completion.
  We will consider sharing raw data and samples collected in the trial to facilitate further research and validation.
Supporting Information: Study Protocol, SAP
Time Frame: We plan to share the primary results within 6 months after the trial ends so that other investigators can understand the results of the trial.
Access Criteria: We plan to share the findings of the trial through journal publications, conference presentations, or other appropriate channels of scientific communication.
  We will consider establishing mechanisms for sharing data and samples, such as data sharing platforms or collaborating with other research teams to share data and samples.